CLINICAL TRIAL: NCT06349759
Title: Randomized, Placebo-Controlled, Double-Masked Study of the Safety and Efficacy of POS (0.75% Phentolamine Ophthalmic Solution) in Subjects Who Have Previously Had Keratorefractive Surgery and Have Decreased Visual Acuity Under Mesopic Conditions
Brief Title: Safety and Efficacy of 0.75% Phentolamine Ophthalmic Solution in Subjects With Post-refractive Surgery Visual Disturbances
Acronym: LYNX-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ocuphire Pharma, Inc. (Industry)
Collaborators: Viatris Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPI-NYXDLD-302 (LYNX-2)
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Mesopic Vision; Night Vision Loss
Keywords: Low light vision
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 0.75% phentolamine ophthalmic solution (Active Comparator): Daily dosing
  Interventions: Drug: phentolamine ophthalmic solution 0.75%, a non-selective alpha-1 and alpha-2 adrenergic antagonist
- phentolamine ophthalmic solution vehicle (Placebo Comparator): Daily dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: phentolamine ophthalmic solution 0.75%, a non-selective alpha-1 and alpha-2 adrenergic antagonist — Once daily dosing
  Other Names: Nyxol
  Arms: 0.75% phentolamine ophthalmic solution
Drug: Placebo — Once daily dosing
  Other Names: phentolamine ophthalmic solution vehicle
  Arms: phentolamine ophthalmic solution vehicle

SUMMARY:
Safety and efficacy of 0.75% Phentolamine Ophthalmic Solution to improve mesopic low contrast visual acuity in subjects with post-refractive surgery visual disturbances.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, double-masked study of the safety and efficacy of POS (0.75% Phentolamine Ophthalmic Solution) in subjects who have previously had keratorefractive surgery and have decreased visual acuity (VA) under mesopic conditions

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 18 years of age
2. Previous history of refractive surgery (eg, PRK, LASIK, SMILE, and RK) and have subject-reported night vision disturbances (eg, glare, halos, and/or starbursts). Symptoms must have been first noted within 2 months following refractive surgery
3. Able to independently comply with all protocol-mandated procedures and to attend all scheduled office visits
4. Able and willing to give written consent to participate in this study
5. Able to self-administer study medication

   Inclusion criteria #6, #7, and #8 must all be met in the same eye:
6. PD ≥ 5 mm under mesopic conditions in at least 1 eye. This test may be repeated once, following an additional 5 min of dark adaptation to the mesopic light conditions if the initial results do not meet this criterion
7. mLCVA ≤ 30 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (20/63 Snellen or worse) in at least 1 eye using the Precision Vision Illuminator Cabinet with 5% translucent contrast chart and a mesopic filter at 4 m
8. ≥ 10 ETDRS letters improvement in mLCVA in at least 1 eye during illumination of the contralateral eye with a Brightness Acuity Tester (BAT) system on the low setting using the Precision Vision Illuminator Cabinet with 5% translucent contrast chart and a mesopic filter at 4 m

Exclusion Criteria:

Ophthalmic (in either eye):

1. Prior unresolved dry eye diagnosis, taking prescription drops for dry eye, or taking artificial tear drops routinely for dry eye
2. Prior history of fluctuating vision
3. Clinically significant ocular disease as deemed by the Investigator (eg, untreated visually significant cataract, glaucoma, corneal edema, uveitis, severe keratoconjunctivitis sicca, retina degeneration, loss of visual field due to glaucoma or stroke, branch retinal vein occlusion, retina flare) that might interfere with the study
4. History or presence of corneal endothelial dystrophy (eg, Fuchs' dystrophy or presence of guttae)
5. Known hypersensitivity to any topical alpha-adrenoceptor antagonists
6. Known allergy or contraindication to any component of the vehicle formulation
7. History of cauterization of the punctum or punctal plug (silicone or collagen) insertion or removal
8. Pseudophakic subjects with extended depth-of-focus or multifocal intraocular lenses (IOLs)
9. Ocular trauma, ocular surgery (eg, IOLs), or laser procedure (eg, LASIK, PRK, SMILE, and RK) within 6 months prior to Screening
10. Use of any topical prescription or over-the-counter (OTC) ophthalmic medications of any kind (including artificial tear drops) within 7 days prior to Screening until study completion, with the exception of lid scrubs with OTC products (eg, OCuSOFT® lid scrub, SteriLid®, baby shampoo, etc.)
11. Recent or current evidence of ocular infection or inflammation (such as current evidence of clinically significant blepharitis, conjunctivitis, or a history of herpes simplex or herpes zoster keratitis at Screening). Subjects must be symptom free for at least 7 days prior to Screening
12. History of diabetic retinopathy, diabetic macular edema, or dry or wet macular degeneration
13. History of any traumatic (surgical or nonsurgical) or nontraumatic condition affecting the pupil or iris (eg, irregularly shaped pupil, neurogenic pupil disorder, iris atrophy, iridotomy, iridectomy, etc.)
14. Unwilling or unable to discontinue use of contact lenses at least 1 hour prior to Screening for soft contact lenses or at least 8 hours prior to Screening for hard gas-permeable contact lenses, and at least 8 hours (for both types of lenses) prior to all other office visits
15. Previously undiagnosed dry eye, at the determination of the Investigator. Dry eye diagnosis should be based on one of the following dry eye test results: tear break-up time < 5 seconds, or corneal fluorescein staining ≥ Grade 2 in the inferior zone or ≥ Grade 1 in the central zone using the National Eye Institute scale

    Systemic:
16. Known hypersensitivity or contraindication to alpha- and/or beta-adrenoceptor antagonists (eg, chronic obstructive pulmonary disease or bronchial asthma; abnormally low BP or HR; second- or third-degree heart blockage or congestive heart failure; or severe diabetes as defined below)

    1. Predisposition to severe hypoglycemia (2 or more serious hypoglycemic episodes requiring assistance within 12 months prior to Screening)
    2. Any hospitalization or emergency room visit due to poor diabetic control within 6 months prior to Screening
    3. Currently untreated diabetes mellitus or previously untreated subjects who initiated oral anti-diabetic medication or insulin within 3 months prior to Screening
    4. Any sign of diabetic retinopathy in either eye
17. Clinically significant systemic disease (eg, severe diabetes as previously defined, myasthenia gravis, cancer, hepatic, renal, endocrine, or cardiovascular disorders) that might interfere with the study
18. Initiation of treatment with or any changes to the current dosage, drug, or regimen of any systemic adrenergic or cholinergic drugs within 7 days prior to Screening or during the study
19. Participation in any investigational study within 30 days prior to Screening or during the study
20. Females of childbearing potential who are pregnant, nursing, planning a pregnancy during the study, or not using a medically acceptable form of birth control. Acceptable methods include the use of at least one of the following: intrauterine device, hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence. A female is considered to be of childbearing potential unless she is 1 year postmenopausal or 3 months post-surgical sterilization. All females of childbearing potential including those post-tubal ligation must have a negative urine pregnancy test result at each visit
21. Resting HR outside 50 to 110 beats per min at Screening. HR may be repeated only once if outside the specified range, following at least a 5-min rest period in the sitting position
22. Hypertension with resting diastolic BP > 105 mmHg or systolic BP > 160 mmHg at Screening. BP may be repeated only once if outside the specified range, following at least a 5-min rest period in the sitting position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects with an increase of at least 15 ETDRS letters read (≥ 3 lines) in the study eye in mLCVA compared to Baseline (Day 1 pre-dose) at Day 15 | Day 15
  To evaluate the efficacy of POS to improve mLCVA in subjects with post-refractive surgery visual disturbances

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pepose, MD, Study Chair — Ocuphire Pharma
Locations (23):
- United States (23):
  - United States Phoenix, Phoenix, Arizona
  - United States Scottsdale, Scottsdale, Arizona
  - United States, Bakersfield, California
  - United States, Glendale, CA, Glendale, California
  - United States, LaJolla, CA, La Jolla, California
  - United States, California, Newport Beach, California
  - United States Rowland Heights, Rowland Heights, California
  - United States Torrance, Torrance, California
  - United States, Jacksonville, FL, Jacksonville, Florida
  - United States Jacksonville, Jacksonville, Florida
  - United States, Tampa, Florida
  - United States Overland Park, Overland Park, Kansas
  - United States Louisville, Louisville, Kentucky
  - United States Fraser, Fraser, Michigan
  - United States Smithtown, Smithtown, New York
  - United States, North Carolina, Garner, North Carolina
  - United States Fargo, Fargo, North Dakota
  - United States, Rhode Island, Warwick, Rhode Island
  - United States, Mt Pleasant, SC, Mt. Pleasant, South Carolina
  - United States Chattanooga, Chattanooga, Tennessee
  - United States Smyrna, Smyrna, Tennessee
  - United States Draper, Draper, Utah
  - United States Lynchburg, Lynchburg, Virginia